CLINICAL TRIAL: NCT04039412
Title: Comparison Between Hybrid, Reverse Hybrid, and Non-Bismuth Levofloxacin Quadruple Regimens for Helicobacter Pylori Infection in Egypt: A Randomized Controlled Trial
Brief Title: Comparison Between Quadruple Regimens for Helicobacter Pylori Infection in Egypt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ayman Magd Eldin Mohammad Sadek (Other Government)
Responsible Party: Sponsor-Investigator, Ayman Magd Eldin Mohammad Sadek, Clinical Professor, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#5089
Record Dates: First submitted 2019-07-04; First posted 2019-07-31 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori Infection; Quadruple Therapy; Egypt

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled (interventional) study conducted at Zagazig University Hospital, internal medicine department clinic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (1) Hybrid regimen (Active Comparator): omeprazole 20mg bid, and amoxicillin 1gm bid in the 1st week, then clarithromycin 500mg bid, omeprazole 20mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid in the 2nd week.
  Interventions: Drug: Hybrid regimen
- (2) Reverse hybrid regimen (Active Comparator): clarithromycin 500mg bid, omeprazole 20mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid for 1 week, followed by omeprazole 20mg bid, and amoxicillin 1gm bid in the 2nd week.
  Interventions: Drug: Reverse hybrid regimen
- (3) Levofloxacin quadruple regimen (Active Comparator): levofloxacin 250mg QD, omeprazole 40mg QD, nitazoxanide 500mg bid, and doxycycline 100mg QD for 10 days. (LOAD)
  Interventions: Drug: Levofloxacin quadruple regimen

INTERVENTIONS:
Drug: Hybrid regimen — two-step (dual-quadruple) treatment
  Arms: (1) Hybrid regimen
Drug: Reverse hybrid regimen — one-step two-phase (quadruple-dual) treatment
  Arms: (2) Reverse hybrid regimen
Drug: Levofloxacin quadruple regimen — non-Clarithromycin non-Bismuth quadruple therapy
  Arms: (3) Levofloxacin quadruple regimen

SUMMARY:
The overall prevalence of H. Pylori in the developing countries is 50.8%, with the highest one presented in Africa (79.1%). Hybrid therapy is supposed to be more effective as a first-line regimen for Helicobacter pylori infection in Egypt than the Reverse hybrid and non-bismuth Levofloxacin quadruple therapies. We are aiming here to compare the Hybrid, Reverse hybrid, and Levofloxacin quadruple therapies as first-line therapy, trying to reach the safest, cost-effective, and compliance-inducing regimen in Egypt. We will conduct a randomized controlled (interventional) study at Zagazig University Hospital, internal medicine department clinic, on 330 patients. 110 patients will be allocated to each regimen.

DETAILED DESCRIPTION:
Introduction:

Although the decreasing prevalence of Helicobacter Pylori (H. Pylori) worldwide, it remains high in developing countries. According to the most recent studies, the overall prevalence of H. Pylori in the developing countries is 50.8%, with the highest one presented in Africa (79.1%).

Unfortunately, the data on the prevalence of H. Pylori, are not available from all the countries of Africa. There is a paucity of information about the magnitude of the problem in Egypt, according to the few available studies, the prevalence is ranging from 71.7-91.7%.

The importance of H. Pylori infection lies in the major role in chronic gastritis, gastric ulcer, and duodenal ulcer, up to gastric adenocarcinoma, and gastric mucosa-associated lymphoid tissue lymphoma.

Diagnosis of H. Pylori can be through invasive tests, which are cumbersome and expensive despite their high sensitivity and specificity. On the contrary, there are more easily and cheaper non-invasive tests, especially H. Pylori stool antigen and urea breath test that has a higher sensitivity than serology.

The decreasing eradication rate of the standard triple therapy (STT) below 80% due to the emergence of resistant strains to Clarithromycin, raise the need for newer therapies that provide higher efficacy, and in the same time, better safety and compliance.

Bismuth-containing quadruple therapy came as the treatment of choice that avoids Clarithromycin use, but it was a non-reasonable option for the countries that are lacking in bismuth salts and/or tetracycline, beside of the complex administration and low safety. It raises the era of the competing sequential and concomitant non-bismuth (clarithromycin containing) quadruple treatments.

A novel two-step (dual-quadruple) treatment called the hybrid therapy (HT), which is actually a combined sequential and concomitant therapy, with a lower cost and better efficacy.

However, the adding of two drugs in the last seven days of the therapy may confuse the patient, making him less willing to complete the treatment that promote the idea of reversing the sequence (quadruple-dual) in what is called the reverse hybrid therapy (RHT), to simplify the treatment in one-step two-phase treatment.

Another non-Clarithromycin non-Bismuth quadruple therapy that is less complex and safer than bismuth quadruple therapy, which is called Levofloxacin quadruple therapy that contains levofloxacin, omeprazole, nitazoxanide, and doxycycline (LOND), showed promising results on the level of the cure rate and low drug resistance profile.

Methods:

Technical Design:

A) The site of study:

The study was conducted in Internal medicine department clinic in Zagazig University Hospitals.

B) Sample size:

Assuming that the eradication rate in patients receiving Hybrid therapy is 91% versus 78.3% in Reverse Hybrid therapy. So, the sample size is 309, using OPEN EPI at power 80% and C.I 95%.

Tools of data collection:

1. Medical history to all participants.
2. Complete clinical examination.
3. The fecal antigen test (FAT) which identifies H. pylori antigen in the stool by enzyme immunoassay was positive in all participants.

Operational design:

A) This is a randomized (interventional) study conducted at Zagazig University Hospital, internal medicine department clinic after informed consent. All the participants were positive for H. pylori fecal antigen test.

B) Steps of performance: (330) participants were chosen from the Internal Medicine Department clinic, grouped into 3 groups:

1. Group 1: (110) participants received reverse hybrid regimen in the form of clarithromycin 500mg bid, omeprazole 20 mg bid, amoxicillin 1gm bid, and metronidazole 500 mg tid for 1 week, followed by omeprazole 20 mg bid, and amoxicillin 1gm bid in the 2nd week.
2. Group2: (110) participants received hybrid regimen in the form of omeprazole 20 mg bid, and amoxicillin 1gm bid in the 1st week, then clarithromycin 500mg bid, omeprazole 20 mg bid, amoxicillin 1gm bid, and metronidazole 500 mg tid in the 2nd week.
3. Group3: (110) participants received Levofloxacin quadruple regimen (LOAD) in the form of nitazoxanide 500 mg bid, levofloxacin 250 mg QD, omeprazole 40 mg QD, and doxycycline 100 mg QD for 10 days

C) Retesting by The fecal antigen test (FAT) after stopping the regimen by at least one month and withholding proton pump inhibitors for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Positive Helicobacter pylori antigen in the stool
* Treatment-naive

Exclusion Criteria:

* Previous treatment for Helicobacter pylori
* Drug hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman MM Sadek, MD, Study Director — Zagazig University
Locations (1):
- Faculty of Human Medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After study publication

REFERENCES:
- [Background] Torres J, Perez-Perez G, Goodman KJ, Atherton JC, Gold BD, Harris PR, la Garza AM, Guarner J, Munoz O. A comprehensive review of the natural history of Helicobacter pylori infection in children. Arch Med Res. 2000 Sep-Oct;31(5):431-69. doi: 10.1016/s0188-4409(00)00099-0. PMID 11179581
- [Background] Zamani M, Ebrahimtabar F, Zamani V, Miller WH, Alizadeh-Navaei R, Shokri-Shirvani J, Derakhshan MH. Systematic review with meta-analysis: the worldwide prevalence of Helicobacter pylori infection. Aliment Pharmacol Ther. 2018 Apr;47(7):868-876. doi: 10.1111/apt.14561. Epub 2018 Feb 12. PMID 29430669
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] El Dine SS, Mubarak M, Salama R, El Raziky M, El Sherbiny E, Zakaria S, Zakaria MS. Low Seroprevalence of anti-CagA antibodies inspite of high seroprevalence of anti-H. Pylori antibodies in rural Egyptian community. Research Journal of Medicine and Medical Sciences. 2008; 3(2):118-23.
- [Background] Diab M, El-Dine SS, Aboul-Fadl L, Shemis M, Omran Z, Badawi A, El-Ghannam M, El-Ray A, Fam N, El-Defrawy I, El-Sherbini E. Helicobacterpylori cag pathogenicity island genes among dyspeptic patients with chronic gastritis. Egypt J Med Microbiol. 2009; 18:43-53.
- [Background] Suerbaum S, Michetti P. Helicobacter pylori infection. N Engl J Med. 2002 Oct 10;347(15):1175-86. doi: 10.1056/NEJMra020542. No abstract available. PMID 12374879
- [Background] Garza-Gonzalez E, Perez-Perez GI, Maldonado-Garza HJ, Bosques-Padilla FJ. A review of Helicobacter pylori diagnosis, treatment, and methods to detect eradication. World J Gastroenterol. 2014 Feb 14;20(6):1438-49. doi: 10.3748/wjg.v20.i6.1438. PMID 24587620
- [Background] Huang YK, Wu MC, Wang SS, Kuo CH, Lee YC, Chang LL, Wang TH, Chen YH, Wang WM, Wu DC, Kuo FC. Lansoprazole-based sequential and concomitant therapy for the first-line Helicobacter pylori eradication. J Dig Dis. 2012 Apr;13(4):232-8. doi: 10.1111/j.1751-2980.2012.00575.x. PMID 22435509
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Georgopoulos SD, Papastergiou V, Karatapanis S. Helicobacter pylori Eradication Therapies in the Era of Increasing Antibiotic Resistance: A Paradigm Shift to Improved Efficacy. Gastroenterol Res Pract. 2012;2012:757926. doi: 10.1155/2012/757926. Epub 2012 Jun 19. PMID 22778723
- [Background] Liou JM, Fang YJ, Chen CC, Bair MJ, Chang CY, Lee YC, Chen MJ, Chen CC, Tseng CH, Hsu YC, Lee JY, Yang TH, Luo JC, Chang CC, Chen CY, Chen PY, Shun CT, Hsu WF, Hu WH, Chen YN, Sheu BS, Lin JT, Wu JY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Concomitant, bismuth quadruple, and 14-day triple therapy in the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2016 Nov 12;388(10058):2355-2365. doi: 10.1016/S0140-6736(16)31409-X. Epub 2016 Oct 18. PMID 27769562
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Liatsos C, Georgopoulos SD. Helicobacter pylori best treatment approach: should a national consensus be the best consensus? Ann Gastroenterol. 2017;30(6):704-706. doi: 10.20524/aog.2017.0183. Epub 2017 Aug 2. No abstract available. PMID 29118570
- [Background] Hsu PI, Tsay FW, Graham DY, Tsai TJ, Tsai KW, Kao JY, Peng NJ, Kuo CH, Kao SS, Wang HM, Lin TF, Wu DC; Taiwan Acid-related Disease (TARD) Study Group. Equivalent Efficacies of Reverse Hybrid and Bismuth Quadruple Therapies in Eradication of Helicobacter pylori Infection in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Sep;16(9):1427-1433. doi: 10.1016/j.cgh.2018.03.031. Epub 2018 Mar 31. PMID 29609070
- [Background] Basu PP, Rayapudi K, Pacana T, Shah NJ, Krishnaswamy N, Flynn M. A randomized study comparing levofloxacin, omeprazole, nitazoxanide, and doxycycline versus triple therapy for the eradication of Helicobacter pylori. Am J Gastroenterol. 2011 Nov;106(11):1970-5. doi: 10.1038/ajg.2011.306. Epub 2011 Oct 11. PMID 21989146
- [Background] Abd-Elsalam S, Kobtan A, El-Kalla F, Elkhalawany W, Nawasany SE, Saif SA, Yousef M, Ali LA, Soliman S, Mansour L, Habba E, Soliman H, Rizk F, Shehata MA. A 2-week Nitazoxanide-based quadruple treatment as a rescue therapy for Helicobacter pylori eradication: A single center experience. Medicine (Baltimore). 2016 Jun;95(24):e3879. doi: 10.1097/MD.0000000000003879. PMID 27310977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted an interventional randomized trial at the internal medicine department clinic, Zagazig University Hospital, Zagazig, Egypt, in the period from July 2018 to June 2019. We allocated the participants attending the clinic by simple randomization over the three treatment groups.
Groups:
- (1) Reverse Hybrid Regimen: clarithromycin 500mg bid, omeprazole 20mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid for 1 week, followed by omeprazole 20mg bid, and amoxicillin 1gm bid in the 2nd week.
  Reverse hybrid regimen: one-step two-phase (quadruple-dual) treatment
- (2) Hybrid Regimen: omeprazole 20mg bid, and amoxicillin 1gm bid in the 1st week, then clarithromycin 500mg bid, omeprazole 20mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid in the 2nd week.
  Hybrid regimen: two-step (dual-quadruple) treatment
Period: Overall Study
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen
Started | 110 | 110 | 110
Completed | 109 | 107 | 108
Not Completed | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen | Total
Number analyzed (Participants) | 110 | 110 | 110 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.05 (9.772) | 32.31 (9.409) | 32.44 (9.713) | 32.27 (9.604)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 55 | 170
  Male | 53 | 52 | 55 | 160
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 110 | 110 | 110 | 330

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Helicobacter Pylori Infection Cure
Description: Measuring the curative rate of each regimen by a fecal antigen test
Time Frame: 40-44 days
Measure: Count of Participants; unit: Participants
Groups:
- (1) Reverse Hybrid Regimen: clarithromycin 500mg bid, omeprazole 20 mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid for 1 week, followed by omeprazole 20 mg bid, and amoxicillin 1gm bid in the 2nd week
- (2) Hybrid Regimen: omeprazole 20 mg bid, and amoxicillin 1gm bid in the 1st week, then clarithromycin 500mg bid, omeprazole 20 mg bid, amoxicillin 1gm bid, and metronidazole 500mg tid in the 2nd week
- (3) Levofloxacin Quadruple Regimen: levofloxacin 250mg QD, omeprazole 40mg QD, nitazoxanide 500mg bid, and doxycycline 100mg QD for 10 days
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen
Number analyzed (Participants) | 110 | 110 | 110
Participants | 102 | 101 | 91

2. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Questionnaire to measure the number of Participants with Treatment-Emergent Adverse Events
Time Frame: 10-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen
Number analyzed (Participants) | 110 | 110 | 110
Participants | 49 | 58 | 44

3. Secondary Outcome: Rate of Helicobacter Pylori Treatment Completion
Description: Questionnaire to evaluate the compliance with each treatment regimen
Time Frame: 10-14 days
Measure: Count of Participants; unit: Participants
Groups:
- (1) Reverse Hybrid Regimen: 109 participants in per-protocol analysis (99.1%)
- (2) Hybrid Regimen: 107 participants in per-protocol analysis (97.3%)
- (3) Levofloxacin Quadruple Regimen: 108 participants in per-protocol analysis (98.2%)
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen
Number analyzed (Participants) | 110 | 110 | 110
Participants | 109 | 107 | 108

ADVERSE EVENTS:
Time Frame: We followed up the occurrence of adverse events after one week of therapy, at the end of treatment, and Up to 45 days.
Description: We divided the severity of adverse event according to the extent of daily activities limitation, into mild, moderate, and severe (no limitation, partial limitation, and profound limitation respectively).
Arm/Group | (1) Reverse Hybrid Regimen | (2) Hybrid Regimen | (3) Levofloxacin Quadruple Regimen
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/107 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/107 | 0/108
Other Adverse Events (participants affected / at risk) | 49/110 | 58/110 | 44/110
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (1) Reverse Hybrid Regimen (N=110) | (2) Hybrid Regimen (N=110) | (3) Levofloxacin Quadruple Regimen (N=110)
Gastrointestinal symptoms (Gastrointestinal disorders) | 41 (41) | 50 (50) | 37 (37)
General symptoms (General disorders) | 8 (8) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04039412/Prot_SAP_000.pdf